CLINICAL TRIAL: NCT07072663
Title: Glymphatic Function and White Matter Integrity in Cerebral Venous Disorders: A Prospective Cohort Study
Brief Title: Glymphatic Function and White Matter Integrity in Cerebral Venous Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: LYS[2025]216-002
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Venous Sinus Thrombosis
Keywords: cerebral venous sinus thrombosis; cerebral venous sinus stenosis; glymphatic system; white matter integrity
MeSH Terms: interventions — BaseLine dental cement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In this study, blood and/or cerebrospinal fluid (CSF) samples will be collected from participants. Prior to collection, informed consent should be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HC group: Sex- and age-matched healthy controls (HCs) without cerebral venous sinus thrombosis (CVST), cerebral venous sinus stenosis (CVSS), or moderate-to-severe intracranial/extracranial arterial stenosis.
  Interventions: Other: Baseline
- CVSS group: Subjects aged ≥18 years with confirmed cerebral venous sinus stenosis (CVSS) exclusively involving the transverse sinus and/or sigmoid sinus (stenosis ≥50%), with or without concomitant internal jugular vein stenosis.
  Interventions: Other: Baseline and 3-month follow-up
- CVST group: Subjects aged ≥18 years with confirmed acute/subacute cerebral venous sinus thrombosis (CVST) (time from onset to diagnosis ≤28 days), with or without concomitant internal jugular vein thrombosis.
  Interventions: Other: Baseline and 3-month follow-up

INTERVENTIONS:
Other: Baseline and 3-month follow-up — At baseline and day 90 (±14) post-enrollment:
  1. Collect clinical data;
  2. Administer multiple scales to assess clinical symptom severity and neuropsychological status;
  3. Perform cranial diffusion tensor imaging (DTI) to evaluate glymphatic function and white matter integrity;
  4. Collect peripheral blood and cerebrospinal fluid (CSF) samples for biomarker level analysis.
  Groups: CVSS group; CVST group
Other: Baseline — At baseline:
  1. Collect clinical data;
  2. Assess intracranial and extracranial arterial and venous systems;
  3. Administer multiple scales to assess neuropsychological status;
  4. Perform cranial diffusion tensor imaging (DTI) to evaluate glymphatic function and white matter integrity;
  5. Collect peripheral blood samples for biomarker level analysis.
  Groups: HC group

SUMMARY:
Cerebral venous disorders, including cerebral venous sinus stenosis (CVSS) and cerebral venous sinus thrombosis (CVST), can obstruct venous blood drainage, leading to intracranial hypertension. However, their effects on glymphatic function and white matter integrity in the brain remain poorly understood.

Therefore, this study will enroll healthy controls, CVSS patients, and CVST patients to compare differences in glymphatic function and white matter microstructural integrity. Additionally, CVSS and CVST patients will undergo a 3-month follow-up to investigate the interrelationships and longitudinal changes among clinical parameters, glymphatic function, and white matter integrity.

DETAILED DESCRIPTION:
Previously, researchers widely believed that the brain lacked a dedicated lymphatic system for clearing metabolic byproducts and wastes. However, recent studies have confirmed the existence of the glymphatic system along perivascular spaces (PVS), which plays a crucial role in metabolic waste clearance, nutrient and neuroactive substance exchange, regulation of central immune responses, and maintenance of cerebral fluid homeostasis. Emerging evidence suggests that dilated draining veins, elevated venous pressure, and increased intracranial pressure may impede glymphatic flow. Consequently, downstream venous pressure alterations-such as local stenosis or thrombosis in cerebral venous sinuses and/or internal jugular veins-could affect parenchymal venule pressure and volume, thereby influencing glymphatic system dynamics.

Preserved myelin integrity is essential for maintaining synchronized and efficient interregional neural communication. Demyelination compromises brain network integration. Diffusion tensor imaging (DTI), an advanced magnetic resonance imaging (MRI) technique for assessing white matter microstructure, can sensitively detect integrity changes. Our preliminary studies identified characteristic bilateral symmetrical cloudy white matter alterations in patients with cerebral venous sinus stenosis, predominantly in periventricular and centrum semiovale regions. However, the precise pathological mechanism remains unclear, and direct evidence linking these changes to chronic venous outflow obstruction is lacking. Although similar imaging findings have not been reported in cerebral venous thrombosis patients, DTI may reveal early microstructural damage, suggesting potential pathological connections.

White matter tracts serve not only as anatomical pathways for glymphatic flow but also depend on glymphatic clearance for metabolic homeostasis. This establishes a bidirectional regulatory relationship: glymphatic dysfunction may induce white matter injury, while white matter lesions could exacerbate glymphatic obstruction. Research indicates that glymphatic impairment may closely correlate with declining white matter integrity, with both potentially forming a mutually reinforcing feedback loop in disease progression across multiple pathologies.

Therefore, this prospective cohort study aims to systematically evaluate glymphatic function and white matter integrity in cerebral venous diseases (including cerebral venous sinus stenosis and thrombosis), further exploring multidimensional correlations among clinical parameters, glymphatic activity, and white matter integrity. The findings may elucidate potential mechanisms of venous-related neural injury.

ELIGIBILITY:
1. Subjects with Cerebral Venous Sinus Stenosis

   Inclusion Criteria:
   * Age ≥18 years, any gender;
   * Definite diagnosis of cerebral venous sinus stenosis confirmed by clinical and imaging examinations;
   * Stenosis limited to the transverse sinus and/or sigmoid sinus, presenting as moderate to severe localized stenosis or occlusion (stenosis degree ≥50%), with or without internal jugular vein stenosis;
   * The subject or their legal representative signs a written informed consent form.

   Exclusion Criteria:
   * Simple anatomical variation or physiological narrowing of the cerebral venous sinus/internal jugular vein without definitive evidence of localized stenosis;
   * Complicated by cerebral venous sinus/cortical vein/internal jugular vein thrombosis;
   * Prior receipt of endovascular treatment for cerebral venous sinus/internal jugular vein, ventricular puncture drainage, or lumbar cistern drainage before enrollment;
   * Presence of moderate to severe stenosis (≥50%) in intracranial or extracranial arteries;
   * History of cerebral infarction, cerebral hemorrhage, or neurosurgery;
   * Complicated by other neurological structural abnormalities such as cerebral small vessel disease, intracranial vascular malformation, dural arteriovenous fistula, intracranial infection, intracranial space-occupying lesion, severe cerebral atrophy, or hydrocephalus;
   * Presence of other diseases affecting glymphatic function (e.g., multiple sclerosis, neuromyelitis optica spectrum disorders, systemic lupus erythematosus, obstructive sleep apnea-hypopnea syndrome, Parkinson's disease, or Alzheimer's disease);
   * Contraindications to MRI (e.g., metal implants, claustrophobia, etc.) or allergy to gadolinium-based contrast agents;
   * Other conditions deemed unsuitable for enrollment by the investigator.
2. Subjects with Cerebral Venous Sinus Thrombosis

   Inclusion Criteria:
   * Age ≥18 years, any gender;
   * Definite diagnosis of acute or subacute phase (onset to diagnosis ≤28 days) cerebral venous sinus thrombosis, with or without internal jugular vein thrombosis, confirmed by clinical and imaging examinations;
   * The subject or their legal representative signs a written informed consent form.

   Exclusion Criteria:
   * Isolated cortical vein thrombosis or isolated cavernous sinus thrombosis;
   * Recurrent intracranial venous sinus thrombosis;
   * Complicated by venous cerebral infarction;
   * Prior receipt of endovascular treatment for cerebral venous sinus/internal jugular vein, ventricular puncture drainage, or lumbar cistern drainage before enrollment;
   * Presence of moderate to severe stenosis (≥50%) in intracranial or extracranial arteries;
   * History of cerebral infarction, cerebral hemorrhage, or neurosurgery;
   * Complicated by other neurological structural abnormalities such as cerebral small vessel disease, intracranial vascular malformation, dural arteriovenous fistula, intracranial infection, intracranial space-occupying lesion, severe cerebral atrophy, or hydrocephalus;
   * Presence of other diseases affecting glymphatic function (e.g., multiple sclerosis, neuromyelitis optica spectrum disorders, systemic lupus erythematosus, obstructive sleep apnea-hypopnea syndrome, Parkinson's disease, or Alzheimer's disease);
   * Presence of severe impaired consciousness, hearing impairment, or aphasia preventing cooperation with examinations or assessments;
   * Contraindications to MRI (e.g., metal implants, claustrophobia, etc.) or allergy to gadolinium-based contrast agents;
   * Other conditions deemed unsuitable for enrollment by the investigator.
3. Healthy Control Subjects:

Inclusion Criteria:

* Gender and age-matched;
* No central nervous system diseases;
* Normal scores on the HAMD-24, HAMA-14, MMSE, MoCA, and PSQI scales;
* No cerebral venous sinus thrombosis, cerebral venous sinus stenosis, or moderate to severe intracranial/extracranial arterial stenosis;
* No contraindications to MRI (e.g., metal implants, claustrophobia, etc.);
* The subject or their legal representative signs a written informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with cerebral venous sinus stenosis (CVSS) and cerebral venous sinus thrombosis (CVST) will be recruited from the outpatient clinic or inpatient wards of the Department of Neurology at Xuanwu Hospital, Capital Medical University, while healthy controls will be recruited from health examination centers or the community.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in DTI-ALPS index from baseline | day 90 (±14) post-enrollment
  The DTI-ALPS (Diffusion Tensor Imaging-Analysis along Perivascular Spaces) index is an imaging biomarker that quantitatively evaluates the function of the brain's glymphatic system using diffusion tensor imaging (DTI) technology, with lower values indicating impaired glymphatic clearance.

SECONDARY OUTCOMES:
Change in PVS score from baseline | day 90 (±14) post-enrollment
  Perivascular spaces (PVS) in the basal ganglia (BG) and centrum semiovale (CSO) are visually scored as: 0 = none, 1 = 1-10, 2 = 11-20, 3 = 21-40, and 4 = >40 on the axial slice with the highest burden and hemicerebrum with higher burden. An increase in PVS score implies a decrease in glymphatic function.
Change in PVS count from baseline | day 90 (±14) post-enrollment
  The number of PVS in the whole brain will be automatically calculated using deep learning algorithms. An increase in PVS count implies a decrease in glymphatic function.
Change in PVS volume from baseline | day 90 (±14) post-enrollment
  The volume of PVS in the whole brain will be automatically calculated using deep learning algorithms. An increase in PVS volume implies a decrease in glymphatic function.
Change in CPV from baseline | day 90 (±14) post-enrollment
  The choroid plexus volume (CPV) will be automatically segmented and calculated using Freesurfer software. An increase in CPV implies a decrease in glymphatic function.
Change in FA from baseline | day 90 (±14) post-enrollment
  Fractional anisotropy (FA) is obtained by Diffusion Tensor Imaging (DTI), and decreased FA values indicate white matter damage.
Change in MD from baseline | day 90 (±14) post-enrollment
  Mean diffusivity (MD) is obtained by Diffusion Tensor Imaging (DTI), and increased MD values indicate white matter damage.
Change in RD from baseline | day 90 (±14) post-enrollment
  Radial diffusivity (RD) is obtained by Diffusion Tensor Imaging (DTI), and increased RD values indicate white matter damage.
Change in AD from baseline | day 90 (±14) post-enrollment
  Axial diffusivity (AD) is obtained by Diffusion Tensor Imaging (DTI), and increased RD values indicate white matter damage.
Change in headache VAS score from baseline | day 90 (±14) post-enrollment
  The visual analogue scale (VAS) for headache assesses pain intensity on a 0-10 scale, where higher scores correlate with greater headache severity.
Change in HIT-6 score from baseline | day 90 (±14) post-enrollment
  Headache Impact Test-6 (HIT-6) is used to assess the comprehensive impact of headaches on quality of life, with total scores ranging from 36 to 78 points. Higher scores indicate greater disruption to daily functioning.
Change in tinnitus VAS score from baseline | day 90 (±14) post-enrollment
  The visual analogue scale (VAS) for tinnitus assesses symptom severity on a 0-10 scale, where higher scores indicate more severe tinnitus.
Change in THI score from baseline | day 90 (±14) post-enrollment
  The tinnitus handicap inventory (THI) is used to evaluate the impact of tinnitus on quality of life, with total scores ranging from 0 to 100. Higher scores reflect more severe disruption to daily functioning.
Change in head noise VAS score from baseline | day 90 (±14) post-enrollment
  The visual analogue scale (VAS) for head noise assesses symptom severity on a 0-10 scale, where higher scores indicate more severe head noise.
Change in HNHI score from baseline | day 90 (±14) post-enrollment
  Head noise handicap inventory (HNHI) is adapted from the tinnitus handicap inventory (THI) by systematically replacing "tinnitus" with "head noise" to evaluate the impact of head noise on quality of life. Total scores range from 0-100, with higher values reflecting more severe functional impairment.
Change in mRS score from baseline | day 90 (±14) post-enrollment
  Modified Rankin Scale (mRS) is used to assess neurological functional recovery status, with total scores ranging from 0 to 6. Higher scores indicate more severe neurological impairment and worse independent living capacity.
Change in HAMD-24 score from baseline | day 90 (±14) post-enrollment
  The 24-item Hamilton Depression Rating Scale (HAMD-24) is used to quantitatively assess the severity of depressive symptoms, with total scores ranging from 0 to 76. Higher scores indicate more severe depression.
Change in HAMA-14 score from baseline | day 90 (±14) post-enrollment
  The 14-item Hamilton Anxiety Rating Scale (HAMA-14) is used to quantitatively assess the severity of anxiety symptoms, with total scores ranging from 0 to 56. Higher scores indicate more severe anxiety.
Change in MMSE score from baseline | day 90 (±14) post-enrollment
  The Mini-Mental State Examination (MMSE) is used to assess cognitive function, with total scores ranging from 0 to 30. Lower scores indicate more severe cognitive impairment.
Change in MoCA score from baseline | day 90 (±14) post-enrollment
  The Montreal Cognitive Assessment (MoCA) is used to assess cognitive function, with total scores ranging from 0 to 30. Lower scores indicate more severe cognitive impairment.
Change in PSQI score from baseline | day 90 (±14) post-enrollment
  The Pittsburgh Sleep Quality Index (PSQI) is used to assess sleep quality, with total scores ranging from 0 to 21 points. A score >5 points indicates sleep disturbance.
Change in fundus parameters from baseline | day 90 (±14) post-enrollment
  Fundus parameters include modified Frisen grading of the fundus, optic disc height, optic nerve sheath width, average retinal nerve fiber layer (RNFL) thickness, etc. These parameters to some extent reflect the degree of intracranial pressure.
Change in lumbar puncture opening pressure from baseline | day 90 (±14) post-enrollment
  The normal lumbar puncture opening pressure range for adults is 70-180 mmH₂O. A pressure >200 mmH₂O typically indicates elevated intracranial pressure.
Change in Farb score from baseline | day 90 (±14) post-enrollment
  The Farb Score is used to evaluate the degree of venous sinus stenosis in subjects with cerebral venous sinus stenosis. The total score ranges from 0 to 8 points, with lower scores indicating higher degrees of stenosis.
Change in thrombus burden from baseline | day 90 (±14) post-enrollment
  The thrombus burden is measured semi-automatically using ITK-SNAP software on contrast-enhanced black-blood thrombus imaging of the head and neck veins.
Venous sinus recanalization rate | day 90 (±14) post-enrollment
  A three-tier classification based on contrast-enhanced MRV of the head and neck is used to evaluate venous sinus recanalization.
Change in biomarker levels in blood and cerebrospinal fluid from baseline | day 90 (±14) post-enrollment
  Blood and cerebrospinal fluid biomarkers include AQP4, Glial Fibrillary Acidic Protein (GFAP), Neurofilament Light Chain (NfL), Aβ40/42, total tau protein (Tau), phosphorylated tau181 (p-Tau181), interleukin (IL)-1β, IL-6, IL-8, IL-10, and tumor necrosis factor (TNF-α).
Incidence of adverse events | day 90 (±14) post-enrollment
  Adverse events included bleeding complications, major bleeding complications (hemoglobin drop ≥19 g/L), symptomatic intracranial hemorrhage, among others.
All-cause mortality | day 90 (±14) post-enrollment
  All-cause mortality refers to deaths from any cause within a studied population, regardless of the specific reason.

CONTACTS AND LOCATIONS:
Overall Officials: Da Zhou, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No